CLINICAL TRIAL: NCT05300477
Title: Augmentation of Medical Readiness and Physical Performance at High Altitude Using Pharmacological Countermeasures
Brief Title: Pharmacological Countermeasures for High Altitude
Status: Active, not recruiting | Phase: Phase 4 | Type: Interventional
Sponsor: United States Army Research Institute of Environmental Medicine (U.S. Federal Agency)
Collaborators: University of Puget Sound (Other)
Responsible Party: Principal Investigator, Roy Salgado, Principal Investigator, United States Army Research Institute of Environmental Medicine
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Other
Other Study IDs: 21-06HC (M-10910)
Record Dates: First submitted 2022-03-17; First posted 2022-03-29 (Actual); Last update posted 2025-03-26 (Actual); Status verified 2025-03

CONDITIONS: Hypobaric Hypoxia
MeSH Terms: interventions — Acetazolamide; Erythropoietin; Epoetin Alfa

STUDY DESIGN:
Intervention Model Description: This study will use a double-blind randomized study design in which one group will receive erythropoietin and the other group will receive the placebo for 4 weeks. After the 4 weeks, both groups will receive acetazolamide.
Who Masked: Participant, Investigator
Masking Description: Participants and Investigators will be blinded to who receives erythropoietin and placebo. Medical providers and a subset of staff will be aware of participants receiving erythropoietin and placebo. Participants, Investigators, and Medical Providers will all be aware of participants administered acetazolamide.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Acetazolamide (Experimental): Acetazolamide (orally) 250 mg twice a day for 3 1/2 days.
  Interventions: Drug: Acetazolamide
- Erythropoietin and Acetazolamide (Experimental): Erythropoietin (subcutaneously) 50 IU /kg three times a week for 4 weeks. After the 4 week Erythropoietin, acetazolamide (orally) 250 mg twice a day for 3 1/2 days.
  Interventions: Drug: Acetazolamide; Drug: Erythropoietin

INTERVENTIONS:
Drug: Acetazolamide — Carbonic Anhydrase Inhibitor
  Other Names: Diamox
Drug: Erythropoietin — Hormone for red blood cell
  Other Names: Procrit
  Arms: Erythropoietin and Acetazolamide

SUMMARY:
The aim of this randomized, double-blind study is to determine whether erythropoietin (Procrit) and acetazolamide: 1) mitigates altitude-induced decrements in performance at moderate altitude (3,000 m) and 2) mitigates altitude-induced decrements in performance and reduce acute mountain sickness during prolonged exposure to high altitude (4,300 m; 15 days). Volunteers will complete 5 study phases: Phase 1) sea level baseline testing and a moderate altitude exposure; Phase 2) 4 week study intervention - randomly assigned to receive erythropoietin or placebo); Phase 3) 3 1/2 days of acetazolamide and a moderate altitude exposure; Phase 4) high altitude acclimatization - 15 days at Pikes Peak; and Phase 5) two week deacclimatization. Test battery include VO2peak, 3.2 km treadmill time trial, measures of gas exchange and ventilation during rest and exercise, and blood collection.

DETAILED DESCRIPTION:
This study will use a double-blind randomized study design in which one group will receive erythropoietin and the other a placebo (saline) for 4 weeks, then both groups will receive acetazolamide. Eighteen men and women volunteers will complete 5 study phases: Phase 1) two week sea level baseline testing (orientation, two VO2peak assessments, three 3.2 km treadmill time-trial, assessment of resting ventilation, venipuncture and capillary blood collection, and Hbmass assessment), and a VO2peak and 3.2 km treadmill time-trial moderate altitude (3,000 m); Phase 2) 4 week intervention to receive subcutaneously erythropoietin or placebo. The erythropoietin (Procrit) dosing regimen will consist of 50 IU/kg three times a week (M-W-F); Phase 3) a second moderate altitude exposure (VO2peak and 3.2 km treadmill time-trial with acetazolamide administered (orally; 250 mg b.i.d) for 3 1/2 nights starting the day before the altitude exposure; Phase 4) high altitude acclimatization in which volunteers will reside for 15 days at 4,300 m altitude (Pikes Peak, Colorado Springs) completing multiple VO2peak assessments and 3.2 km treadmill time-trials, resting ventilation, venipuncture and capillary blood collection; and Phase 5) deacclimatization phase to assess changes in hematological biomarkers after returning from Pikes Peak. This study consists of 41 visits over a ~10 week time period. Visits will take place in Natick, MA and the Pikes Peak High Altitude Research Laboratory at Colorado Springs. Additional assessments that will be completed multiple times during the study include: acute mountain sickness questionnaire, lung gas diffusion at rest and during exercise, oxygen saturation, arterialized blood gases (PO2, PCO2, pH, HCO3) and heart rate during rest, exercise, and sleep, and muscle tissue oxygenation. The primary outcome is 3.2 km treadmill time-trial performance. Secondary outcomes include: incidence and severity of acute mountain sickness, ventilation and gas exchange, Hbmass, Hb concentration, Hct, arterialized blood gases, lung diffusion at rest and during exercise, oxygen saturation and heart rate during rest, exercise, and sleep.

ELIGIBILITY:
Inclusion Criteria:

* Age 18-40 years
* In good health as determined by the Office of Medical Support & Oversight (OMSO) General Medical Clearance
* Runs at least 3 times per week and able to complete a two mile run in ≤ 21 minutes (Civilian Volunteers) or passed his/her most recent Army Combat Fitness Test (ACFT) (Military Volunteers Only)
* Willing to not exercise, or drink alcoholic and/or caffeinated beverages 24 hours prior to each testing session or the acute altitude exposure to 3,000 m
* Abstain from alcoholic beverages during the 15 day residence at the summit of Pikes Peak
* Abstain from drinking alcohol or caffeine at least 24 hours before a testing session during Phases 1 and 3
* Willing to stay and exercise in an altitude chamber (the size of a dorm room) for ~2.5 hours
* Wiling to reside at the summit of Pikes Peak (4,300 m altitude) and share dormitory area (bunk area, shower, and bathroom), potentially with people of the opposite sex for 15 days
* Up to date on COVID-19 vaccination

Exclusion Criteria:

* Women who are pregnant or planning to become pregnant during the study
* Taking prescription medication, or over-the-counter medications other than contraceptives, unless approved by OMSO & PI
* Born at altitudes greater than 2,100 m (7,000 ft)
* Living in areas that are more than 1,200 m (4,000 ft) or have traveled to areas that are more than 1,200 m for five days or more within the last 2 months
* Prior diagnosis of High Altitude Pulmonary Edema (HAPE) or High Altitude Cerebral Edema (HACE)
* Musculoskeletal injuries that compromise the ability to walk/run on a treadmill or hike steep terrain
* Abnormal blood count in accordance with OMSO - Normal Hb men: 12.6-17.7 g·dL-1 and women: 11.1-15.9 g·dL-1 or Normal Hct men: 37.5-48% and women: 34.0-45%, or presence of abnormal blood chemicals (hemoglobin S or Sickle Cell Trait)
* Any history of malignancy
* Personal or family history of blood clots
* Abnormal prothrombin time/partial thromboplastin time (PT/PTT) test or problems with blood clotting
* History of thromboembolic disease, hypertension, and known risk factors of cardiovascular disease
* Blood donation within 8 weeks of beginning the study
* History of seizures
* History of inflammatory bowel disease
* Any recent (within 4-6 weeks) and or expected history of prolonged periods of immobility or limited activity (including recent or upcoming surgery)
* No evidence of iron deficiency (ferritin < 45 ng/ml)
* Smokers or tobacco/nicotine (unless quit > 1 month prior to study orientation)
* History of asthma
* Experience recent (< 1 month of starting the study) cold, coughs, or respiratory tract infections
* Allergy to skin adhesive
* Known allergy to sulfa drugs
* Evidence of apnea or sleeping disorder
* Present condition of alcoholism, use of anabolic steroids, other substance abuse issues
* Inability to tolerate iron supplement

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 18 (Estimated)
Dates: Start 2022-05-27 (Actual); Primary Completion 2023-09-30 (Actual); Study Completion 2025-09-30 (Estimated)

PRIMARY OUTCOMES:
3.2 km self-paced treadmill time trial performance | 35 minutes
  Time to complete self-paced 3.2 km treadmill time trial (min:sec)

SECONDARY OUTCOMES:
VO2peak | 30 minutes
  Peak aerobic capacity will be assessed using a metabolic cart.
Lake Louise Acute Mountain Sickness Score | 10 minutes
  Acute mountain sickness and severity will be assessed using the Lake Louise acute mountain sickness questionnaire. This Likert scale assess acute mountain sickness with scores ranging from 0 to 12. Zero indicates no acute mountain sickness and 12 indicates severe acute mountain sickness.
Ventilation rate | 20 minutes
  Ventilation rate will be assessed using a pneumotachometer.
Percent body fat | 10 minutes
  Percent body fat will be assessed using Dual Energy X-ray Absorptiometry.
Oxygen Saturation | 35 minutes
  Oxygen saturation will be assessed using a finger pulse oximeter.
Erythropoietin | 4 hours
  Erythropoietin will be assessed using an ELISA.
Hematocrit | 5 minutes
  Hematocrit will be assessed using manual hematocrit method.
Reticulocyte | 2 hours
  Reticulocyte will be assessed using a hematology analyzer.
Ferritin | 2 hours
  Ferritin will be assessed using an ELISA.
C-reactive protein | 2 hours
  C-reactive protein will be assessed using an ELISA.
Soluble transferrin | 2 hours
  Soluble transferrin will be assessed using an ELISA.
Arterialized capillary PO2 | 5 minutes
  Arterialized capillary PO2 will be assessed using a blood gas analyzer.
Arterialized capillary PCO2 | 5 minutes
  Arterialized capillary PCO2 will be assessed using a blood gas analyzer.
Arterialized capillary pH | 5 minutes
  Arterialized capillary pH will be assessed using a blood gas analyzer.
Hbmass | 20 minutes
  Hbmass will be assessed using the CO-rebreathing procedure.
Muscle tissue oxygenation | 35 minutes
  Muscle tissue oxygenation will be assessed using a non-invasive near-infrared spectroscopy.
Lung Diffusion of carbon monoxide | 35 minutes
  Lung Diffusion of carbon monoxide will be assessed using a spirometer.

CONTACTS AND LOCATIONS:
Overall Officials: Roy Salgado, PhD, Principal Investigator — United States Army Research Institute of Environmental Medicine
Locations (1):
- USARIEM, Natick, Massachusetts, United States